CLINICAL TRIAL: NCT01883726
Title: Comparison of Two Nasoalveolar Molding Techniques in Complete Unilateral Cleft Lip Patient
Acronym: NAM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 102-1267C
Record Dates: First submitted 2013-06-03; First posted 2013-06-21 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-04

CONDITIONS: Unilateral Complete Cleft Lip
Keywords: Unilateral complete cleft lip, Nasoalveolar molding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Grayson NAM (Experimental): Intervention: Grayson nasoalveolar molding This technique uses an acrylic plate to mold the alveolar segments and uses an extension to mold the alar cartilage of the nasal component. The construction is made by gradual modification of the acrylic plate with periodic acrylic add on and grinding. When the alveolar gap is reduced to 5 mm, nasal component are added to gradually mold the nasal cartilage and other nasal structures.
  Interventions: Device: Grayson's presurgical nasoalveolar molding
- Figueroa NAM (Experimental): Intervention: Figueroa's nasoalveolar molding Figueroa technique uses labial tapes and acrylic relief to the palatal plate to approximate alveolar gap [3]. The nasal component is added in the beginning of the treatment to mold the nasal cartilage.
  Interventions: Device: Figueroa's presurgical nasoalveolar molding

INTERVENTIONS:
Device: Grayson's presurgical nasoalveolar molding — Grayson NAM
  Arms: Grayson NAM
Device: Figueroa's presurgical nasoalveolar molding — Figueroa NAM
  Arms: Figueroa NAM

SUMMARY:
Two types of Presurgical Nasoalveolar Molding (NAM) coexist in Craniofacial Center in Chang Gung Memorial Hospital. The objective of this study is to compare the number of clinical visits, total prices, complications and nasal symmetry between these two NAM reconstruction methods.

DETAILED DESCRIPTION:
Grayson's NAM reconstruction starts with alveolar molding first. The alveolar molding is made by gradual modification of the acrylic plate with periodic acrylic add on and grinding. After the alveolar cleft gap is less than 5 mm (usually at the end of second months), nasal molding was added to the alveolar molding plate.

Figueroa's NAM reconstruction use labial tapes and acrylic relief to the palatal plate to approximate alveolar gap. The device starts with nasal and alveolar molding simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* Complete unilateral cleft lip infant
* Signed informed consent

Exclusion Criteria:

* Incomplete unilateral cleft lip infant
* Association of other craniofacial anomalies

Ages: 1 Week to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2010-05; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
The nasal morphology - Nostril height 1 | (T1) at initial visit
  Nostril height: the vertical distance between horizontal reference lines to the highest point of nostril aperture.
The nasal morphology - Nostril height 2 | (T2) after nasoalveolar molding (participants' nasoalveolar molding will be finished before surgery, an expected average of 3-months old)
  Nostril height: the vertical distance between horizontal reference lines to the highest point of nostril aperture.
The nasal morphology - - Nostril height 3 | (T3) one week after surgery
  Nostril height: the vertical distance between horizontal reference lines to the highest point of nostril aperture.
The nasal morphology - Nostril height 4 | (T4) 6 months after surgery
  Nostril height: the vertical distance between horizontal reference lines to the highest point of nostril aperture.
The nasal morphology - Nostril width 1 | (T1) at initial visit
  Nostril width: The widest horizontal distance between the inner medial and lateral border of nostril aperture.
The nasal morphology - Nostril width 2 | (T2) after nasoalveolar molding (participants' nasoalveolar molding will be finished before surgery, an expected average of 3-months old)
  Nostril width: The widest horizontal distance between the inner medial and lateral border of nostril aperture.
The nasal morphology - Nostril width 3 | (T3) one week after surgery
  Nostril width: The widest horizontal distance between the inner medial and lateral border of nostril aperture.
The nasal morphology - Nostril width 4 | (T4) 6 months after surgery
  Nostril width: The widest horizontal distance between the inner medial and lateral border of nostril aperture.
The nasal morphology - Nasal sill height 3 | (T3) one week after surgery
  Nasal sill height: the vertical distance between the horizontal reference line to the lowest border of nostril aperture.
The nasal morphology - Nasal sill height 4 | (T4) 6 months after surgery
  Nasal sill height: the vertical distance between the horizontal reference line to the lowest border of nostril aperture.
The nasal morphology - nostril area 1 | (T1) at initial visit
  Nostril area: the area presented by nostril aperture.
The nasal morphology - nostril area 2 | (T2) after nasoalveolar molding (participants' nasoalveolar molding will be finished before surgery, an expected average of 3-months old)
  Nostril area: the area presented by nostril aperture.
The nasal morphology - nostril area 3 | (T3) one week after surgery
  Nostril area: the area presented by nostril aperture.
The nasal morphology - nostril area 4 | (T4) 6 months after surgery
  Nostril area: the area presented by nostril aperture.

SECONDARY OUTCOMES:
duration of NAM | From initial of nasoalveolar molding to finish of nasoalveolar molding (participants' nasoalveolar molding will be finished before surgery, an expected average of 3-months old)
  Duration of NAM = Operation date - NAM initiation date
total number of visits before surgical correction | From the initial visit to the date of surgery (participants' surgery will be performed on 3-month of age)
  Total number of orthodontic visit or NAM adjustment = number of adjustment of NAM
cost of treatment | From initial orthodontic visit to finish of NAM (participants' nasoalveolar molding will be finished before surgery, an expected average of 3-months old)
  Cost = cost of each visit of orthodontic and adjustment of NAM before surgery
NAM complications | From initial of NAM to finish of NAM (participants' nasoalveolar molding will be finished before surgery, an expected average of 3-months old)
  Any complication like mucosa ulceration and facial skin irritation

CONTACTS AND LOCATIONS:
Locations (1):
- Chun-Shin, Chang, Taipei, Taiwan, Taiwan

REFERENCES:
- [Derived] Chang FC, Huang JJ, Wallace CG, Hsiao YC, Chen ZC, Liao YF, Chen PK. Comparison of Facial Growth between Two Nasoalveolar Molding Techniques in Patients with Unilateral Complete Cleft Lip. Plast Reconstr Surg. 2023 Nov 1;152(5):1078-1083. doi: 10.1097/PRS.0000000000010448. Epub 2023 Mar 21. PMID 36940137
- [Derived] Chang CS, Wallace CG, Pai BC, Chiu YT, Hsieh YJ, Chen IJ, Liao YF, Liou EJ, Chen PK. Comparison of two nasoalveolar molding techniques in unilateral complete cleft lip patients: a randomized, prospective, single-blind trial to compare nasal outcomes. Plast Reconstr Surg. 2014 Aug;134(2):275-282. doi: 10.1097/PRS.0000000000000361. PMID 24732649